CLINICAL TRIAL: NCT03954691
Title: Targeting Potassium Channels to Reprogram Glioblastoma Microenvironment: in Vitro and in Vivo Studies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Cristina Limatola, Principal Investigator, Neuromed IRCCS
Other Study IDs: RF-2018-12366215
Record Dates: First submitted 2019-05-11; First posted 2019-05-17 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — glioblastoma biopsies
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: brain tumor-immune cells communication — tumoral and immune cell isolation from biopsis

SUMMARY:
The investigators want to verify the hypothesis that targeting the calcium-activated (KCa3.1) and the voltage-dependent K channel (Kv1.3) could be a valuable therapeutic strategy to reprogram cells of the innate immune system, with the aim to fight glioma, a deadly CNS tumor. The investigators will use murine models of glioma, injecting GL261 cells in the brain of syngeneic C57BL6 mice, to study the effect of K channel inhibition on the activation of microglia (M), macrophages (Mf) and NK cells. The investigators will use M and vesicles released from these cells, re-educated toward an anti-tumor phenotype, to interfere with the vicious circle responsible of uncontrolled tumor growth and will study the role of NK cells in tumor-M/Mf communication. The investigators will also investigate how K channels interfere with the communication of innate immune cells and brain cells like neurons and astrocytes, with experiments focused on synaptic transmission and calcium imaging, investigating the effect of modulation of the tumor microenvironment.

DETAILED DESCRIPTION:
Specific Aim 1:

Specific Aim 3:

To investigate whether M, or Mf-derived micro-vesicles, delivered to the brain of mouse bearing glioma could affect glioma growth and mice survival. This will allow to better define the role of M in controlling glioma growth as a function of its activation state and of KCa3.1 and Kv1.3 channel expression and activity. OBJECTIVE: from this aim the investigators expect to verify whether brain delivery of differently polarized M (or M-derived vesicles), or M/Mf, could represent a meaningful approach to counteract glioma growth and to lengthen mice survival.

Investigate the relationship between CD11b+ and NK cells upon KCa3.1 and Kv1.3 inhibition or NK cell depletion. OBJECTIVE: data obtained will help to understand whether the activation state of M/Mf affects NK cell accumulation in the tumor site and their cytotoxic activity, whether NK cells modulate M/Mf activation, with effects on tumor growth, and the eventual role played by K+ channels. Our preliminary data showing that TRAM-34 treatment increased the mRNA level of IL-15 in the brain of glioma-bearing mice (FIG3) would suggest an IL-15-mediated increased accumulation of NK cells in the tumor region, similarly to previous evidence (19).

To investigate the roles of KCa3.1 and Kv1.3 channels in the interaction between glioma and the surrounding parenchyma. OBJECTIVE: to identify possible mechanisms of altered communication in the brain of mice treated with K+ channel inhibitors by studying K+ currents, excitatory and inhibitory synaptic transmission and astrocytes activation state, under normal and hypoxic conditions (corresponding to different position in the tumor mass). Altered expression and function of ion channels in glioma cells isolated from mice treated with functionally different M and M-derived vesicles will also be investigated.

Experimental Design Aim 1:

Experimental Design Aim 2:

Experimental Design Aim 3:

This will be investigated with M polarized in culture, treated with TRAM-34 or PAP-1, silenced by siRNA specific for KCa3.1 (9) or isolated from KCa3.1-/- or Kv1.3 -/- mice and transplanted in the brain of glioma bearing mice by brain injection or intranasal delivery. Brain injection of M will be performed similarly to glioma injection (21). Intranasal (i.n.) cell application will be performed during a short isoflurane anesthesia. Before treatment, all animals will receive 100 U hyaluronidase i.n. dissolved in 12 µL of sterile PBS and one hour later a microglia suspension (3 × 105 in 12 µL of sterile PBS) or vehicle (PBS) will be applied using the same procedure. Microglia application will be repeated every 3 days until mice sacrifice. To check for M delivery in brain tumor region, control experiments will be performed using GFP-labeled M, obtained from sibling CX3CR1GFP/+ mice, already available in our laboratory. To prepare micro-vesicles, M will be treated with ATP (1mM) for 30 min (20). Different centrifugation steps will be performed and the homogeneity of vesicle dimension will be evaluated in parallel experiments by dynamic light scattering. Fixed volumes of this preparation (4microL) will be administrated intra nasally every 3 days until mice sacrifice. M and Mf-derived micro-vesicle-transplanted mice will then be analyzed for tumor volume and mice survival investigated as described (9).

This will be performed on cells isolated (by human biopsy and mice brain) by FACS sorting or by magnetic separator (CD11b+ cells), and assayed in vitro for phagocytic and cytotoxic activity. The investigators will also perform analysis of gene expression and electrophysiological recordings (patch clamp) of ion channel function on M and on tumor cells in vitro and ex vivo in brain slices. These experiments will be performed in TRAM-34 or PAP-1 treated or in KCa3.1-/- or KV1.3-/- glioma bearing mice. M/Mf-NK cell interaction will be also studied looking at NK-induced M/Mf alteration and M/Mf-induced NK alteration. At this aim the investigators will deplete NK cell population with repeated injection of anti NK1.1 antibody in glioma bearing mice, to analyze the activation state of M/Mf cell population.

For this aim the investigators will use electrophysiological, fluorescence and confocal microscope analysis in acute brain slice preparations. A detailed description of the functional role of microglial K+ channels in modulating glioma progression will be provided. In particular, the functional properties of KCa3.1 and Kv1.3 channels expressed by microglial cells in control and glioma injected mice will be evaluated in acute brain slices by means of the patch-clamp techniques. The effects of K channel blockade on neuronal signaling and on astrocytes reactivity will be also evaluated in the same conditions. Fluorescence-based digital Ca2+ imaging will be used to assess the role of these channels in microglial [Ca2+]i regulation. Using electrophysiological measurements, in combination with immunochemical, PCR, siRNA analysis, the investigators will also analyze the modulation of K channels in glioma. Using acute brain slices from glioma-injected mice, the investigators will also assess whether treatment of mice with polarized M affects the expression and function of glioma ion channels known to contribute to the transformed phenotype, such as KCa3.1 channels, BK channels, and volume-activated Cl channels. These experiments will be performed in hypoxic and non-hypoxic areas of the tumor, identified ex post by evaluating the HIF-1alfa expression.

Methodologies and statistical analyses: The iterative method of "Camussi et al." (20) will be followed. The investigators will use the following relation where n is the number of animals: n>2sigma^2 (z alpha/D)^2. As an example, to estimate the number of mice necessary to obtain a significance alpha=0.09, a difference D in treatment effect on a given parameter, the investigators need to know the standard deviation sigma. Since sigma^2 is unknown, it must be substituted with an estimate of sampling variance s^2. If the investigators give to s^2=0.01, the investigators have that n>18, so the investigators predict to use 20 mice per experimental group. Our experience with mice suggests that it is a reasonable number. Statistical significance will be assessed by one-way ANOVA for parametrical data, as indicated; "Holm-Sidak" test will be used as post-hoc test; "Mann and Withney" test for non-parametrical data. Where appropriate, Student's t-test or analysis of variance (ANOVA) will be used.

ELIGIBILITY:
Inclusion Criteria:

- glioma patients who undergo neurosurgery

Exclusion Criteria:

- biopsies from patients with brain tumor different than glioma

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: glioma patients who undergo neurosurgery for glioblastoma surgical eradication
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
glioblastoma cells | 6 months
  observational studies on cells isolated from tumor specimens

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Cristina Limatola, Pozzilli, Is
  - Cristina Limatola, Pozzilli